CLINICAL TRIAL: NCT05027555
Title: Effect of Multisensory Training on Gait Variability in People With Parkinson's Disease
Brief Title: Multisensory Training in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21MMHIS153e
Record Dates: First submitted 2021-08-21; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
Keywords: Multisensory training; Gait variability
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multisensory training group (Experimental): The intervention is a 50-minute session and 2-sessions/week, totaling 6 weeks
  Interventions: Other: Multisensory training
- Conventional training group. (Active Comparator): The intervention is a 50-minute session and 2-sessions/week, totaling 6 weeks
  Interventions: Other: Conventional training

INTERVENTIONS:
Other: Multisensory training — Multisensory training included marching on the foam with visual deprivation and treadmill training with visual deprivation
  Arms: Multisensory training group
Other: Conventional training — Conventional training included strengthening, balance training and gait training
  Arms: Conventional training group.

SUMMARY:
People with Parkinson's disease (PD) were characterized by many motor symptoms, including rigidity, postural instability, bradykinesia, and resting tremor. These motor symptoms might cause gait dysfunction. Gait dysfunction represented a common sign of PD, including reduced gait velocity, reduced stride length, reduced arm swing, and increased gait variability. Poor postural control in people with PD might result to increase gait variability and then increase fall risk. Previous studies reported that proprioceptive-vestibular multisensory training improved postural stability in people with PD. However, no literature investigated the effects of proprioceptive-vestibular multisensory training on gait variability. Therefore, the purpose of this study is to examine the effect of proprioceptive-vestibular multisensory training on gait variability in people with PD.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD
* Hoehn and Yahr stage I to III
* Age 60~80 y/o
* Mini-Mental State Examination (MMSE) ≥24
* Ability to ambulate independently (with or without walking aid)

Exclusion Criteria:

* Affecting the peripheral vestibular system
* Medical condition that substantially influenced their gait and balance performance
* People had joined any rehabilitation past 1 month

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait variability | Change from baseline at 6 weeks
  Using GAITRite system to measure coefficient of variation

SECONDARY OUTCOMES:
Gait performance | Change from baseline at 6 weeks
  Using the GAITRite system to evaluate saptiotemporal parameters
Sensory organization test | Change from baseline at 6 weeks
  Using NeuroCom Smart Balance Master
Timed up and go test | Change from baseline at 6 weeks
  To evaluate functional mobility
Dynamic Gait Index | Change from baseline at 6 weeks
  To evaluate functional mobility

IPD SHARING:
Plan to Share IPD: Undecided